CLINICAL TRIAL: NCT01967654
Title: Implementing Tobacco Use Guidelines in Community Health Centers in Vietnam
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-00413
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Technical assistance, training, plus clinical reminder system (Experimental): To assess the contextual factors of the intervention settings (district level policies and organizational level characteristics) that may influence tobacco use treatment in CHCs and to inform additional modifications to the proposed implementation strategies.
  Interventions: Other: Technical Assistance, training and clinical reminders
- TTC + referral to community health workers (Experimental): To compare the effectiveness and cost effectiveness of two multi component implementation strategies.
  Interventions: Other: Referral to Community Health Worker

INTERVENTIONS:
Other: Technical Assistance, training and clinical reminders
  Arms: Technical assistance, training, plus clinical reminder system
Other: Referral to Community Health Worker
  Arms: TTC + referral to community health workers

SUMMARY:
Vietnam has a smoking prevalence that is the second highest among South East Asian countries (SEACs). With a population of approximately 90 million, Vietnam also has the second largest total number of adult smokers (over 16 million) in SEA. According to the World Health Organization (WHO), most reductions in mortality from tobacco use in the near future will be achieved through helping current users quit. Tobacco use treatment, as defined by the U.S. Preventive Health Service Guideline (Guideline) on Treating Tobacco use and Dependence, is evidence-based and highly cost-effective. Yet, in the U.S. and globally, adoption of recommended care is suboptimal. The objective of this proposal is to fill the current research-to-practice gap by conducting a randomized controlled trial that compares the effectiveness and cost effectiveness of two practical and highly replicable strategies for implementing evidence-based guidelines for the treatment of tobacco use in public health clinics in Vietnam. The proposed implementation strategies draw on evidence-based approaches, and the WHO's recently released guidelines for implementing Article 14 of the Framework Convention on Tobacco Control (FCTC). The FCTC is an evidence-based treaty that was developed by the WHO in response to the globalization of the tobacco epidemic. Vietnam ratified the FCTC in 2004; however, they have not taken steps to implement Article 14 which specifies the need to integrate best practices for treating tobacco use and dependence into routine preventive care. The proposed implementation strategies also build on the growing literature that supports the effectiveness of integrating community health workers as members of the health care team to improve access to preventive services.

DETAILED DESCRIPTION:
Aim 1: To conduct a formative evaluation.

The formative evaluation has three components: 1) Key informant interviews with leaders in the public health sector responsible for developing and implementing policy in Vietnam to assess contextual factors (e.g. district level policies) that may influence implementation and dissemination; 2) Focus groups with current smokers to inform adaptations to the current training curriculum and counseling manual; and 3) baseline study site assessments to assess organizational readiness to change and current policies and practices to inform necessary adaptations to the proposed system changes.The investigators will develop semi-structured interview and focus group guides and adapt survey tools guided by the conceptual model described above as well as a robust literature on factors that influence implementation and dissemination.

Data collection. 1) Key informant interviews. The investigators will conduct key informant interviews with at least one senior level staff person from the following stakeholder groups: a) MOH central level agencies involved in tobacco control such as VINACOSH, and the Ministries of Education and Training and Science and Technology; b) Executive Directors of the Vietnam Medical Association and the Vietnam Public Health Association; c) WHO Vietnam; d) at the provincial level, a representative from the Department of Health and Preventive Medicine Center; and e) four district health directors in the two target provinces (HaNoi and Thai Nguyen) for a total of about 16 interviews. The investigators use a semi-structured interview guide organized by constructs found to influence implementation and dissemination outcomes.52-56 These include external factors (tobacco control policies, national priorities for resource allocation and relative priority of tobacco control, relative priority of smoking cessation) perceived barriers to implementing guideline recommended cessation services, perceived commitment of leadership in and outside the MOH, perceived challenges to maintaining and disseminating changes in service delivery at the local and province level. Recruitment for key informant interviews: Using a purposive sampling approach, ISMS will leverage their contacts to assist in recruiting stakeholders for the key informant interviews through email invitations to participate. Research staff will then follow-up by telephone to enroll stakeholders in the study. The investigators will conduct these interviews. 2) Focus groups: An experienced facilitator from ISMS will conduct six focus groups (3 in each study district) with current smokers (6-8 participants, 4 male and 2 female groups). The focus groups will assess expectations about health benefits of quitting, past cessation history, including availability, affordability and use of cessation medications, knowledge of cessation resources, and attitudes towards the proposed intervention. There is a relatively large database on the knowledge and attitudes about tobacco use among smokers in Vietnam. Therefore, the groups will focus more on access to treatment, attitudes towards pharmacotherapy and treatment preferences. Inclusion/exclusion criteria include: current smoker (smoked in past 7 days), patient of a CHC in one of the two study districts, and age 18 and over. Recruitment for focus groups: the same methods as were used to recruit patients to the pilot study. Patients will be screened for current tobacco use in the CHCs, asked to participate if they meet eligibility criteria and given a date and time for the meeting. Consent will be obtained at the time of the focus group. 3) Baseline study site assessments: In all enrolled study sites the following will be conducted: a) an assessment of baseline organizational characteristics. This includes data on setting-level variables shown to influence the implementation of practice guidelines including number of FTE staff, clinic volume, policies and systems. A a practice environment checklist will be used to inventory current policies, workflow, systems (e.g. chart systems) and staff roles and responsibilities in general, and specifically related to tobacco use treatment. b)Semi-structured interviews with clinical and administrative key informants (clinical director, 2 CHWs and 3 providers per site) to supplement the checklist data and to elaborate on potential barriers and facilitators for tobacco use treatment. c) A provider and CHW survey (tested in the pilot research and based on a survey from the WHO that was validated in Vietnamese). Surveys will assess baseline knowledge, attitudes and current practice patterns related to tobacco use treatment to inform additional modifications in training materials. d) Organizational readiness to change: provider surveys will include the Change Process Capability Questionnaire(CPCQ), a validated tool that is applicable to primary care practice.

AIM 2: To compare the effectiveness and cost effectiveness of two implementation strategies to increase adherence to tobacco use treatment guidelines, and AIM 3: To explore organizational factors hypothesized to influence the relationship between the implementation strategies and implementation effectiveness. The Aims will be combined for the remainder of the Approach section because of overlaps in design and data collection.

A two arm, randomized trial comparing approach will be used: ARM 1) technical assistance, training, and clinical reminder system (TTC), and ARM 2) TTC+ referral to a CHW for additional counseling and follow-up. The investigators will conduct a baseline assessment of provider adherence to tobacco use treatment by collecting patient exit interviews (PEIs) (i.e., surveys conducted immediately after the patient visit) from 50 patients per site who meet eligibility criteria as current smokers. We will then implement the components of ARM 1 and 2. At 12 months post implementation we will conduct PEIs with another 50 smokers per site. These patients will be asked to consent to follow-up surveys at 3 and 6 months to assess smoking abstinence.

Study Site eligibility and recruitment. The investigators have chosen two provinces to represent both an urban and rural setting. Thai Nguyen and Hanoi The district we have selected in Hanoi is representative of those CHCs located in the central part of the city and the district in Thai Nguyen is representative of the rural CHCs in that province. Site criteria include having at least one physician, >4 allied health care professional staff, >5 CHWs and a patient population of at least 4000. Using methods for site recruitment used by ISMS, the Director of the District Health Centers will introduce our study to all CHCs that fit these criteria through a letter of introduction and follow-up telephone or in person contacts. Among those expressing interest, we will randomly select 26 CHCs (13 rural and 13 urban). Sites will be randomly assigned in a 1:1 ratio to the intervention conditions within urban and rural strata. We will recruit sites in 3 successive waves.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligibility:
* Current patients at community health center for routine visit
* 18 years or older
* Current or regular smoker (>1 cigarette in past 7 days)
* Willingness to complete survey
* Provider eligibility:
* Provider at community health center
* 18 years or older
* Willingness to complete survey or interview

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Adherence to tobacco use treatment guidelines | 4-6 weeks
  To assess the primary outcome of provider adherence to tobacco treatment guidelines, the investigators will conduct patient exit interviews (PEI) (surveys conducted immediately after the patient visit) with 50 smokers pre and 50 postimplementation at each site (1300 in each study period).

SECONDARY OUTCOMES:
Smoking abstinence | 6 months
  Using accepted standards for measuring cessation outcomes, all patients who complete a PEI in the post intervention period will be followed prospectively to assess 3 and 6 month 7-day point prevalence abstinence, defined as any smoking (even a puff) in the past 7 days. Surveys will be conducted in person and smoking abstinence will be validated using carbon monoxide (CO) monitoring with abstinence defined as a CO<10ppm.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shelley, MD, MPH, Principal Investigator — NYU School of Medicine
Locations (1):
- Institute of Social and Medical Studies, Hanoi, Vietnam

REFERENCES:
- [Derived] Shelley D, Cleland CM, Nguyen T, VanDevanter N, Siman N, Van Minh H, Nguyen N. Effectiveness of a Multicomponent Strategy for Implementing Guidelines for Treating Tobacco Use in Vietnam Commune Health Centers. Nicotine Tob Res. 2022 Feb 1;24(2):196-203. doi: 10.1093/ntr/ntab189. PMID 34543422
- [Derived] Shelley D, VanDevanter N, Cleland CC, Nguyen L, Nguyen N. Implementing tobacco use treatment guidelines in community health centers in Vietnam. Implement Sci. 2015 Oct 9;10:142. doi: 10.1186/s13012-015-0328-8. PMID 26453554